CLINICAL TRIAL: NCT05853003
Title: Neuromuscular Ultrasonography Assessment of Optic Nerve in SLE
Brief Title: Neuromuscular Ultrasonography Assessment of Optic Nerve in Systemic Lupus Eryhematosus
Status: Completed | Type: Observational
Sponsor: Amira M elSonbaty (Other)
Responsible Party: Sponsor-Investigator, Amira M elSonbaty, Amira Elsonbaty, Assiut University
Organization: Assiut University (Other)
Other Study IDs: bending
Record Dates: First submitted 2023-02-19; First posted 2023-05-10 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Optic Neuropathy
MeSH Terms: conditions — Optic Nerve Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
assessing the role of neuromuscular ultrasound in optic nerve involvement in systemic lupus patients.

DETAILED DESCRIPTION:
Evaluating the role of neuromuscular ultrasound in optic nerve involvement in systemic lupus patients.by measuring the diameter of optic nerve at certain site and comparing it to healthy subjects measurements and to asses NMUS ability to detect optic neuropathy in lupus patients in comparison to conventional techniques including opthalmologist evaluation and visual evoked potential

ELIGIBILITY:
Inclusion Criteria:

* Adult
* group of SLE patients, who fulfilled Systemic Lupus International Collaborating Clinics classification criteria for SLE (SLICC) with or without symptoms of optic neuropathy
* another group of apparently healthy subjects with no. history of chronic conditions

Exclusion Criteria:

* Any patient with optic neuritis due to causes other than lupus was excluded from the study: ex.

  * Post traumatic neuropathy
  * Purely degenerative neuropathy
  * Diabetic neuropathy
  * Toxic neuropathy
  * Neuropathies related to infections
  * Drug induced neuropathy e.g: quinine and some antibiotics, ethambutol
  * Infections e.g. measles, mumps, Lyme disease, etc.
  * Other Autoimmune diseases like sarcoidosis, B.D
  * Tumor causing Inc. intracranial tension.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adult SLE patients, who fulfilled Systemic Lupus International Collaborating Clinics classification criteria for SLE (SLICC) and another group of an apparently healthy subjects will be added to the study
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
comparing diameter (in mm2) of optic nerve in SLE patients and compare them to healthy subjects | over 1 year
  comparing diameter (in mm2) of optic nerve in SLE patients and compare them to healthy subjects

CONTACTS AND LOCATIONS:
Overall Officials: Amira elsonbaty, PHD, Principal Investigator — Assiut University
Locations (1):
- Assuit university hospital, Asyut, Egypt